CLINICAL TRIAL: NCT01509326
Title: A Randomized Clinical Trial of Chiropractic Care for Headaches With and Without an Acupressure Device
Brief Title: Chiropractic and Acupressure for Headaches
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: Dr. Zaxx Co. (Unknown)
Responsible Party: Principal Investigator, Howard Vernon, Professor, Canadian Memorial Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112049
Record Dates: First submitted 2012-01-04; First posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Cervicogenic Headache; Tension-type Headache; Migraine Headache
Keywords: headache; chiropractic; manipulation; acupressure; self-care
MeSH Terms: conditions — Post-Traumatic Headache; Tension-Type Headache; Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chiropractic (Active Comparator): spinal manipulation, mobilization, massage, advice, exercises
  Interventions: Other: chiropractic treatment
- Chiropractic PLUS pillow (Experimental): spinal manipulation, mobilization, massage, advice, exercises, pillow
  Interventions: Device: Dr. Zaxx pillow

INTERVENTIONS:
Other: chiropractic treatment — 12 sessions over 4 weeks
  Arms: Chiropractic
Device: Dr. Zaxx pillow — Daily use of an acupressure pillow
  Arms: Chiropractic PLUS pillow

SUMMARY:
This study will investigate the effect of chiropractic treatment with and without the use of an acupressure pillow for cervical headaches. Subjects will be randomly allocated to groups with and without the pillow and will be followed for five weeks. The primary outcome measure will be headache frequency. The investigators predict that the group using the pillow on a daily basis will demonstrate significantly greater decrease in headache frequency over a 5-week interval.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* ages 21-60
* recurrent headaches
* sub-occipital tenderness
* a minimum of 4 headaches per month

Exclusion Criteria:

* migraine with aura
* sinus headache
* any other organic pathology
* any contraindications to cervical manipulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Headache frequency from a Headache Diary | change from baseline in headache frequency at 5 weeks
  Daily Headache Diary

SECONDARY OUTCOMES:
Headache disability | baseline / end of treatment (5 weeks)
  Headache Disability Index
Treatment satisfaction | end of treatment (5 weeks)
  Small scale for rating satisfaction with treatment
Adverse events | up to five weeks
  pain, stiffness, dizziness

CONTACTS AND LOCATIONS:
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada

REFERENCES:
- [Background] Vernon H, Jansz G, Goldsmith CH, McDermaid C. A randomized, placebo-controlled clinical trial of chiropractic and medical prophylactic treatment of adults with tension-type headache: results from a stopped trial. J Manipulative Physiol Ther. 2009 Jun;32(5):344-51. doi: 10.1016/j.jmpt.2009.04.004. PMID 19539116
- See also: Institutional webpage — http://www.cmcc.ca